CLINICAL TRIAL: NCT06644872
Title: The Effect of Short-term Bed Rest on Cardiac Function Measured by Cardiac Magnetic Resonance Imaging
Acronym: MRtime
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Bente Kiens, Professor, University of Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MRTIME
Record Dates: First submitted 2024-10-04; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-06

CONDITIONS: Rest; Healthy
Keywords: Cardiac output; bedrest; Healthy
MeSH Terms: interventions — Bed Rest

STUDY DESIGN:
Intervention Model Description: single-arm repeated measurement study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cardiac magnetic resonance measurements (Experimental): Healthy participants will undergo a three and half-hour experimental day including repeated measurements of cardiac magnetic resonance and blood sampling.
  Interventions: Other: Bedrest

INTERVENTIONS:
Other: Bedrest — Investigation of the effect of short-term bed rest (3 hours) on heart function, measured by cardiac magnetic resonance, in healthy participants ( males and females)

SUMMARY:
The primary objective of this study is to investigate the effect of short-term bed rest (4 hours) on heart function, measured by cardiac magnetic resonance (CMR), in healthy participants. This aim will be addressed through a single-arm repeated study, assessing participants during three hours of bedrest.

The hypothesis is that short-term bed rest will decrease cardiac output measured by repeated CMR scans.

This study will also investigate the reproducibility of CMR within a narrow time frame. Limited data are available on these aspects, despite their critical importance for conducting consecutive examinations, both in clinical practice and research trials10-12. The study also aims to investigate the appliances of short-time measures of cardiac function.

DETAILED DESCRIPTION:
The study will be conducted as a single-arm repeated measurement study in healthy participants (n=19). The participants will undergo a three and half-hour experimental day.

Initially, potential participants are invited to an information meeting and after informed consent, a control screening of MR contraindications is fulfilled. Following inclusion, the test day are conducted. The participants will arrive after a 4-hour period with no intake of food and drinks, except 250g of water, and by passive transportation (train, bus, or car). After arrival, a vein catheter is inserted into the antecubital vein. Then, a basal venous blood sample (-15 min) is drawn (4 ml in total) for analysis of plasma catecholamine and acetylcholine, and blood pressure is taken. Thereafter, the first basal CMRs will be performed with ECG monitoring.

During the test day, the participants will undergo five 15 min CMR imaging scans at 0, 30, 60, 120 and 180 mins. The first three are consecutive measurements with short breaks between, therefor the participants will lay in the scanner for the first 75 min and stay in bed in between the two sequential measurements. The participants will be in bedrest throughout the experimental day. Venous blood samples (4 ml) are obtained at 75, 110, and 170 min, where also blood pressure is taken. In total, up to 25 ml blood is obtained during the test day. The duration of the test day is 4.5 hour.

The time requirements for each participant are summarized:

* Information meeting and screening, approximately 1.5 hour
* 1 test day of approximately 4.5 hour.

Screening At the screening, height, and body weight will be measured, and a questionnaire on contraindications for CMR will be completed to ensure compliance to the scanner. The daily study leader will ask about previous illnesses, medication intake, alcohol, and smoking habits.

Statistical considerations Measures of myocardial function are highly reproducible when assessed using CMR, and interstudy and cohort coefficients of variation are in the range of 3%-5%10-12. In this study, the primary outcome is change in cardiac output after bed rest compared with the first CMR scanning before bed rest.

In an ongoing study, preliminary observations reveal a decrease of mean±SD -10±9% in CO and -4.1±5.9% in LVEF in both healthy participants and those with heart failure after two hours of bed rest, as evaluated by CMR.

For the upcoming study, the aim is to be able to detect a minimal effect difference of 10% and variation in the CMR data sampling as evident from unpublished observations described above. Sample size calculations were performed, considering a conservative approach with a power of 95% and a significance level of 0.05, utilizing paired Student's t-test for data evaluation. The calculations are as follows:

* For changes in CO, 11 participants would be sufficient to detect a 10% change.
* For changes in LVEF, 19 participants would be adequate to detect a 4% change. To account for potential dropouts or failed scans, the plan is to include, up to 29 participants, until 19 completed experimental days have been obtained .

In regard to the analysis plan, a t-test comparing the first (no bedrest) and the last CMR scan (4h bed rest) is the primary endpoint, further a mixed model will be performed to assess the difference in cardiac function throughout the day.

Participants Participants in this study consist of 19 healthy male and female participants.

ELIGIBILITY:
Inclusion Criteria:

Male or female.

* Age between 18-80 years old.
* No use of medications with influence on heart function.
* For ethical reasons, we only include participants who are willing to be informed on new health information, as CMR may reveal relevant secondary health findings.

Exclusion Criteria:

* Diabetes, kidney, or liver disease.
* Contraindications to CMR, e.g., abdominal height exceed limitations of the MR-scanner, pacemaker, aortastent, neurostimulator, or other electronic device implanted, implanted metal devices, severe claustrophobia, or physiological diseases.
* Pregnant, lactating, or planning to become pregnant within the study period.
* In ongoing cancer treatment.
* Blood donation during and < 1 month prior to study.
* Simultaneous participation in other clinical trials potentially affecting the study outcome.
* Inability, physically or mentally, to comply with the procedure required by the study protocol ad evaluated by the primary investigator, study manager or clinical responsible.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
cardiac output | 0-4 hours
  Change in cardiac output will be measured assessed by repeated cardiac magnetic resonance measurement after shortterm bed rest compared with before bedrest.

SECONDARY OUTCOMES:
Left ventricular ejection fraction | 0-4 hours
  Left ventricular ejection fraction willl be measured by cardiac magnetic resonance before and after shortterm bedrest

CONTACTS AND LOCATIONS:
Overall Officials: Bente Kiens, D.sci, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
a decision has not jet been made